CLINICAL TRIAL: NCT04337463
Title: An Open, Dose-escalation and Expansion Study With a Dual TORC1/2 Inhibitor of ATG-008 Combined With PD-1 Antibody of Toripalimab in Advanced Solid Tumors
Brief Title: ATG-008 Combined With Toripalimab in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Li Zheng, Professor, Sichuan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATG-008-HX-001
Record Dates: First submitted 2020-03-21; First posted 2020-04-07 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATG-008 and Toripalimab (Experimental): Toripalimab will be combined with ATG-008.
  Interventions: Drug: ATG-008; Drug: Toripalimab

INTERVENTIONS:
Drug: ATG-008 — Tablet
Drug: Toripalimab — IV infusion

SUMMARY:
This is an open-label, single-arm study with dose-escalation and expansion phases to access ATG-008 combined with Toripalimab in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Know and voluntarily sign informed consent.
2. Age 18-70 years old (including 18 and 70 years old), weight ≥45 Kg.
3. At least one measurable lesion according to the RECIST 1.1 and RANO evaluation criteria.
4. ECOG performance status score is 0 or 1.
5. Blood chemistry test results, meet the following results:

   1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × normal upper limit (ULN)
   2. Total bilirubin ≤ 1.5 × ULN
   3. Serum albumin> 29 g / L
   4. Creatinine ≤ 1.5 × ULN or 24-hour serum creatinine clearance ≥ 50 mL / min
   5. Lipase and amylase ≤ 2 × ULN.
6. Adequate bone marrow function and meets the following results:

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 109 / L
   2. Platelets ≥ 75 × 10^9 / L
   3. Hemoglobin ≥ 90 g / L.
7. Except for hearing loss and hair loss, all toxicity caused by previous anti-tumor therapy must have returned to ≤ Grade 1 (according to NCI-CTCAE version 5.0).
8. Life expectancy is longer than 3 months.

Exclusion Criteria:

1. Have a history of hepatic encephalopathy.
2. Have a thyroid disorder with a clinically significant thyroid dysfunction judged by the investigator (not applicable for thyroid cancer in dose expansion phase).
3. Active or history of upper gastrointestinal bleeding, ulcers, or esophageal varices with bleeding within 6 months.
4. Have a history of HIV infection and/or acquired immunodeficiency syndrome
5. Major surgery has been performed within 4 weeks before the first dose, or is expected during the study period.
6. Have a history of organ transplantation (eg., liver transplantation).
7. Poorly-controlled pleural or pericardial effusion during the screening period.
8. Other primary malignancies occurred within 5 years before the first administration of the study drug with the exception of locally curable malignancies
9. Suffering from active or previously recurring autoimmune diseases or under such a risk.
10. Systemically immunosuppressive drugs are currently used within 14 days of the first dose.
11. The investigator considers that the complications or other situations of the subject may affect compliance with the protocol, or are not suitable for participation in this study.
12. Subjects with diabetes or glycated hemoglobin (HbA1c)> 7%.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-23 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
MTD | Within 21 days after dosing
  Maximum Tolerated Dose
RP2D | Within 21 days after dosing
  Recommended phase 2 dose
ORR | Through study completion (approximately 2 years)
  Overall Response Rate

SECONDARY OUTCOMES:
Cmax | Day 1 - Day 15
  Peak Plasma Concentration (Cmax)
AUC | Day 1 - Day 15
  Area under the plasma concentration versus time curve (AUC)
DOR | 12 months
  Duration from the first observation of at least PR to time of disease progression, or deaths due to disease progression, whichever occurs first.
DCR | 12 months
  Disease Control Rate (DCR=CBR+Stable Disease[SD; for a minimum of 12 weeks])
PFS | 12 months
  Duration from start of study treatment to PD or death (regardless of cause), whichever comes first
OS | 12 months
  The estimates of Kaplan-Meier

CONTACTS AND LOCATIONS:
Overall Officials: Li Zheng, Principal Investigator — West China Hospital
Locations (2):
- China (2):
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - West China of Sichuan University, Chengdu, Sichuan